CLINICAL TRIAL: NCT03674190
Title: A Study Comparing the Outcome of Anterior Lumbar Fusion and Total Lumbar Disc Replacement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to find patients that accepted the study
Sponsor: Svante Berg (Other)
Collaborators: Yara Asterfjord (Unknown)
Responsible Party: Sponsor-Investigator, Svante Berg, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MollyMoa
Record Dates: First submitted 2018-09-02; First posted 2018-09-17 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Disc Disease Degenerative; Disk Degeneration; Disc Disease Lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease | interventions — Total Disc Replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Lumbar Interbody Fusion (Experimental): Surgical treatment Anterior Lumbar Interbody Fusion
  Interventions: Procedure: Anterior Lumbar Interbody Fusion
- Total disc replacement (Active Comparator): Surgical treatment total disc replacement in the lumbar spine
  Interventions: Procedure: Total Disc Replacement

INTERVENTIONS:
Procedure: Anterior Lumbar Interbody Fusion — Anterior Lumbar Fusion(ALIF)
  Arms: Anterior Lumbar Interbody Fusion
Procedure: Total Disc Replacement — Total Disc Replacement
  Arms: Total disc replacement

SUMMARY:
Total lumbar disc replacement has previously been compared to posterior fusion of the lumbar spine, showing some favor towards total disc replacement. The study aims to compare total disc replacement to anterior fusion, sparing the muscles of the back and thus comparing the two different methods using the same surgical approach.

DETAILED DESCRIPTION:
A total of 170 patients are planned to be enrolled in the study. If the patients meet the inclusion criteria and accept to participate they will be randomized to either anterior lumbar fusion or total disc replacement. The method of choice will be blinded for the patients until the two year follow up is completed.

Follow-up: after one and two years. Questionnairs: ODI, VAS, EuroQol, and GA Flexion- Extension X-ray after one and two years Complications will be retrieved from the patient journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disabling pain from degenerative disc disease(DDD) both clinical and radiological, in one or two segments of the lumbar spine from L4-S1, were prolonged conservative treatment has failed.
* The patient should be able to understand swedish written and spoken.
* The patient should be between the ages 18-65. The patient has to accept to participate in the study

Exclusion Criteria:

* More than two degenerated segments.
* Degeneration above the L4 segment.
* Did not agree to participate in the study
* Previous history of tumor, vertebral fracture, infection, lumbar fusion and dominating leg pain.
* Need for posterior decompression
* Pregnancy
* Psychiatric illness or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
ODI, Oswestry Disability Index | Two years
  ODI questionnaire. ODI (Oswestry disability index, self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel, 0-5 zero indicating the least amount of disability and 5 indicating most severe disability)

SECONDARY OUTCOMES:
VAS, Visual Analogue Scale | Two years
  VAS Scale, VAS (Visual Analogue Scale, 0 no pain, 100 worst possible pain) of back and leg,collected from questionnaires
Segment Mobility | Two years
  Flexion Extension X-ray
Patient reported back pain after two years in Swespine national registry | Two years
  GA (Global Assessment of back pain, patient-based evaluation of leg and back pain as compared to preoperatively,1-5, 1 disappeared and 5 worsened) ,collected from questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Svante Berg, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Spine Center Göteborg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No